CLINICAL TRIAL: NCT06608862
Title: The Impact of Hormonal Contraceptive Use, Body Composition, Muscular Strength and Iron Status on Fracture Risk and Bone Quality in Adult Females from 18-35 Years
Brief Title: The Impact of Hormonal Contraceptive Use and Lifestyle Factors on Fracture Risk and Bone Quality in Young Female Adults
Acronym: FH
Status: Recruiting | Type: Observational
Sponsor: Bundeswehr University Munich (Other)
Responsible Party: Principal Investigator, Annette Schmidt, PhD, Prof. Dr. Annette Schmidt, Bundeswehr University Munich
Other Study IDs: Female Health
Record Dates: First submitted 2024-09-17; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Osteoporosis; Osteopenia; Fracture Reduction; Body Composition; Nutrition; Hemoglobin; Muscle Strength; Bone Density; Contraception Behavior; Physical Activity; Menstrual Irregularities
Keywords: impact of lifestyle factors on bone quality; impact of hormonal contraceptive use on bone quality; impact of body composition on bone quality; impact of nutrition and energy balance on bone quality; impact of amenorrhea on bone quality; impact of physical activity on bone quality; impact of the occupation soldier on bone quality; impact of muscle strength on bone quality
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Contraception Behavior; Motor Activity; Menstruation Disturbances

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — A drop of capillary blood from the fingertip is collected for hemoglobin analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Female soldiers: Female soldiers from the university of the Bundeswehr in Munich, which are all of German nationality and between 18 and 35 years of age.

SUMMARY:
The study on hand is based on a cross-sectional design and aims to acquire 1) descriptive data on the physical state and health condition of female soldiers in the German armed forces. 2) a possible influence of different contraceptive methods as well as physical activity, body composition, strength, nutrition, and hemoglobin levels on bone health should be investigated.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 35 years
* female
* willing to participate under a pseudonym
* occupational soldiers
* free from chronic or acute musculoskeletal injury

Exclusion Criteria:

* for the bioelectrical impedance: electronic implants like defibrillator, pregnancy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study focuses on female soldiers, which are underrepresented in research.
Study Population: Female soldiers between 18-35 years.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
T-Score | Measured at baseline and at 12 months after enrollment
  Changes in bone density T-Scores measured via ultra-sonic

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Bundeswehr Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Anonymous data might be shared, however the German Bundeswehr owns the data by now and has to decide on any data issues.